CLINICAL TRIAL: NCT04861285
Title: Evaluation of Gingival Displacement With RACESTYPTINE Solution and RACEGEL: a Prospective, Comparative Randomized Clinical Trial.
Brief Title: Gingival Displacement With RACESTYPTINE Solution and RACEGEL: a Prospective, Comparative Randomized Clinical Trial.
Acronym: RETRACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Septodont (Industry)
Collaborators: Slb Pharma (Other); Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RETRACT; 2021-A00179-32 (Other: identifier from the French National Agency of Health (ANSM))
Record Dates: First submitted 2021-04-23; First posted 2021-04-27 (Actual); Last update posted 2021-11-29 (Actual); Status verified 2021-06

CONDITIONS: Gingival Retraction Techniques
Keywords: gingival retraction, dental impression

STUDY DESIGN:
Intervention Model Description: Study subject (tooth) will be randomized in a 1:1:1 allocation ratio between the 3 gingival retraction techniques.
Who Masked: Outcomes Assessor
Masking Description: Blinding will be done to the assessors who analyzed dental impression to reduce bias to gingival tissue displacement assessment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- RACESTYPTINE Solution with cord (Experimental): The participant will receive RACESTYPTINE Solution into the sulcus. The solution is used in combination with a non-medicated gingival retraction cord.
  Interventions: Device: RACESTYPTINE Solution with cord
- RACEGEL with cord (Experimental): The participant will receive RACEGEL into the sulcus. The gel is used in combination with a non-medicated gingival retraction cord.
  Interventions: Device: RACEGEL with cord
- RACEGEL without cord (Experimental): The participant will receive RACEGEL into the sulcus. No cord will be added.
  Interventions: Device: RACEGEL without cord

INTERVENTIONS:
Device: RACESTYPTINE Solution with cord — The dentist inserts a non-medicated gingival retraction cord into the sulcus and then impregnates the cord in situ with a few drops of RACESTYPTINE Solution. The impregnated cord is left in place a few minutes and then removed. The gingival sulcus is washed and gently air-dried before taking impression.
  Arms: RACESTYPTINE Solution with cord
Device: RACEGEL with cord — The dentist applies a sufficient amount of RACEGEL directly into the sulcus, following the contour of the prepared tooth, and then inserts a non-medicated gingival retraction cord into the sulcus. The impregnated cord is left in place a few minutes and then removed. The sulcus is washed and gently air-dried before taking impression.
  Arms: RACEGEL with cord
Device: RACEGEL without cord — The dentist applies a sufficient amount of RACEGEL directly into the sulcus, following the contour of the prepared tooth. The gel is left in place a few minutes and then removed. The sulcus is washed and gently air-dried before taking impression.
  Arms: RACEGEL without cord

SUMMARY:
The study design is a prospective, multi-center randomized, controlled, open label, 3-arm parallel group, post market clinical follow-up (PMCF) Clinical Trial.

The aim of the study is to collect clinical performance and safety data from RACEGEL and RACESTYPTINE Solution. Three gingival retraction techniques are being studied: RACESTYPTINE Solution with cord, RACEGEL with cord and RACEGEL without cord.

The study will demonstrate the expected performance of these 3 techniques in terms of sulcus opening, i.e. a lateral gingival displacement of at least 200 µm (state of the art) allowing the realization of pre-prosthetic impression with subgingivally margins. 90 subjects (teeth) requiring a dental restoration with subgingival margins for placement of a fixed prosthesis will be enrolled in 3 groups (30 in each group). For each participant, two dental impressions are performed: one impression before the gingival retraction and one impression immediately after the gingival retraction. Both impressions are scanned with 3D dental scanner and images are superimposed before analysis of tissue displacement.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female (age ≥18 years),
* Patient requiring a dental restoration with subgingival margins on one or more teeth with placement of a single or multiple fixed prosthesis. Partially edentulous patients can be enrolled.
* Good oral hygiene
* Healthy periodontium and gingiva: probing depth ≤3 mm, no evidence of gingival inflammation (gingival index ≤ 1), attachment loss (attached gingival >2 mm), bleeding on probing, or plaque accumulation (plaque index < 3)
* Patient who received information and gave written consent.
* Patient affiliated with a social security/protection plan.

Exclusion Criteria:

* Contraindication to taking impression evidenced at the latest on the day of inclusion visit (gingival index ≥2, sign of attachment loss or tooth mobility, probing depth >3 mm).
* Known allergy to aluminum, aluminum salts or to one of the compounds of the formula of the gingival retraction material, or to one of the compounds of the impression material.
* Patient with an unbalanced systemic disease (diabetes, thyroid disorders, history of oropharyngeal cancer),
* Simultaneous participation in another interventional clinical investigation or trial,
* Vulnerable Subjects

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2021-05-10 (Actual); Primary Completion 2021-11-05 (Actual); Study Completion 2021-11-12 (Actual)

PRIMARY OUTCOMES:
Quantitative assessment of the lateral gingival displacement | Day 0
  Two dental impressions are performed per participant at the same visit : one impression before the gingival retraction and one impression immediately after the gingival retraction. Both impressions are scanned with 3D dental scanner and images are superimposed before analyses. The lateral gingival displacement corresponds to the difference between pre- and post-displacement sulcus width measured in the 2 superimposed images of the pre- and post-retraction scanned models.

SECONDARY OUTCOMES:
Quantitative assessment of the vertical gingival displacement | Day 0
  The vertical gingival displacement corresponds to the greatest vertical distance between the crest of the gingiva in the 2 superimposed images of the pre- and post-retraction scanned models.
Oozing control assessment | Day 0
  The dentist visually assesses the presence or absence of crevicular fluid in the sulcus immediately after removing the retraction material.
Bleeding control assessment | Day 0
  The dentist visually assesses the stop of gingival bleeding (if there was one prior to the gingival retraction step), immediately after removing the retraction material.
Gingival index | Day 0 (before and after the gingival retraction), Day 14 (end of study visit)
  The Gingival Index records gingival inflammation on the prepared tooth in 3 grades according the following criteria:
  Grade 0 = Normal gingiva. Grade 1 = Mild inflammation - slight change in color, slight edema. No bleeding on probing.
  Grade 2 = Moderate inflammation - redness, edema, glazing. Bleeding on probing. Grade 3 = Severe inflammation - marked redness and edema, ulceration. Tendency toward spontaneous bleeding.
Papilla Bleeding index | Day 0 (before and after the gingival retraction), Day 14 (end of study visit)
  The Papilla Bleeding Index assesses gingival inflammation in the interdental papillae by recording bleeding on probing in the interdental areas. A periodontal probe is passed along the gingival margin to provoke bleeding and clinical findings are recorded according the following criteria:
  Grade 0 = No bleeding on probing. Grade 1 = isolated bleeding spots present. Grade 2 = blood forms a red line on gingival margin. Grade 3 = heavy profuse bleeding.
Probing depth | Day 0 (before and after the gingival retraction), Day 14 (end of study visit)
  The probing depth measures the distance (in mm) from the free end of the gingival margin to the bottom of the periodontal pocket with a calibrated periodontal probe. A healthy periodontium and gingiva has a probing depth ≤3 mm. A probing depth >3 mm is pathologic.
Adverse events | Day 0, Day 14 (end of study visit)
  Adverse events clinically observed by the dentist during the gingival retraction and impression procedures (Day 0) and at the end of study visit (Day 14) will be used to assess the safety.

CONTACTS AND LOCATIONS:
Overall Officials: Hugues Colombel, DDS, Principal Investigator — Cabinet dentaire (Rennes)
Locations (5):
- France (5):
  - Cabinet dentaire, Cesson-Sévigné
  - Cabinet dentaire Dr Rubin, Rennes
  - Cabinet dentaire Magister, Rennes
  - Cabinet dentaire, Rennes
  - Cabinet dentaire - Médipole 35, Tinténiac

IPD SHARING:
Plan to Share IPD: No